CLINICAL TRIAL: NCT06795373
Title: A Single-center, Single-arm, Open-label Phase IIA Clinical Trial to Investigate Efficacy and Safety of Ritlecitinib (PF-06651600) in Participants With Chronic Spontaneous Urticaria
Brief Title: Ritlecitinib (PF-06651600) in Participants With Chronic Spontaneous Urticaria
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated study
Sponsor: Ahuva D Cices (Other)
Responsible Party: Sponsor-Investigator, Ahuva D Cices, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-01277
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Chronic Spontaneous Urticaria; CSU
Keywords: Chronic Spontaneous Urticaria; CSU; Ritlecitinib
MeSH Terms: conditions — Chronic Urticaria | interventions — PF-06651600

STUDY DESIGN:
Intervention Model Description: This is a prospective phase IIA study to investigate efficacy, safety, and tolerability of ritlecitinib treatment in participants with persistent, progressive, or recurrent chronic spontaneous urticaria (CSU). It is designed as an open label, single-arm, single-center pilot study. A total of up to 20 participants with a physician-based diagnosis of CSU and the other characteristics mentioned in the inclusion criteria will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- persistent, progressive, or recurrent chronic spontaneous urticaria (CSU). (Experimental): Participants with persistent, progressive, or recurrent chronic spontaneous urticaria (CSU).
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Ritlecitinib — Once daily dose of 100mg of ritlecitinib taken orally for 12 weeks
  Other Names: PF-06651600

SUMMARY:
The purpose of this research study is to see if a drug called ritlecitinib is safe and effective for treating chronic spontaneous urticaria (CSU). CSU is hives and itching lasting over six weeks. Ritlecitinib is approved by the Food and Drug Administration (FDA) to treat another condition, but it is not approved for treating CSU. Participation is expected to last 20 weeks and include 7 clinic visits. This study will involve physical examinations, blood tests, looking at and taking pictures of participant's skin and hives, optional skin biopsies, and hearing tests. Eligible participants for this study will take ritlecitinib for 12 weeks and complete a daily diary about their skin and hives. The main risks of being in this study are side effects from ritlecitinib. Less than 1 in 10 people taking ritlecitinib experience diarrhea, acne, hives, rash, inflammation of hair follicles, dizziness, and increased blood levels of creatine phosphokinase (a muscle protein). Participants could also experience a rare but serious side effect, such as shingles, unusual infection, cancer, or blood clot. Benefits of participating in this study include a potential improvement in participant's condition and quality of life. Participating in this study may also help researchers develop new ways of helping future patients.

ELIGIBILITY:
INCLUSION CRITERIA:

Participants are eligible to be included in the study only if all the following criteria apply:

* Participant has been informed about study procedures and medications and has provided informed consent prior to initiation of any study-specific activities/procedures
* Participant is able to communicate with the investigator, and understands and complies with the requirements of the study
* Age ≥ 18 to ≤ 65 years of age at screening
* Participant has a negative Tuberculin purified protein derivative (PPD) or QuantiFERON TBGold test (QFT) at screening or within the last 12 months.
* Chronic spontaneous urticaria diagnosis ≥ 3 months at the time of screening visit 1
* Diagnosis of CSU inadequately controlled by second-generation H1-antihistamines (sgAH) at enrollment, as defined by the following:

  * The presence of itch and hives for ≥ 6 consecutive weeks at any time prior to screening visit 2 despite current use of an approved dose of H1-antihistamine
  * Urticaria Activity Score over 7 days (UAS7) (range 0-42) ≥ 16 and Hive Severity Score over 7 days (HSS7) (range 0-21) ≥ 8 during the 7 days prior to enrollment
* Participant must have been on or failed a sgAH at approved or increased doses (up to 2 or 4x the approved dose) for treatment of CSU prior to the Baseline visit and must have documented current use on the day of screening visit ○ If participants are currently on a sgAH, they must continue the same dose throughout the trial

EXCLUSION CRITERIA:

Disease Related

* Urticaria is solely due to inducible urticaria
* Active dermatologic diseases (or conditions) other than chronic urticaria, with urticaria wheals or angioedema symptoms such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary or acquired angioedema (eg, due to C1 inhibitor deficiency)
* Any other active skin disease associated with chronic itching that might influence, in the investigator's opinion, the study evaluations and results (eg, atopic dermatitis, dermatitis herpetiformis, senile pruritus, etc.)

Other Medical Conditions

* History of, or a concurrent, clinically significant illness, medical condition or laboratory abnormality that, in the investigator's opinion, could affect the conduct of the study
* Active immunosuppression by previous (5 x half-lives or 12 weeks, whichever is longer) or current systemic cytotoxic therapies
* Uncontrolled current illness, including, but not limited to the following: Ongoing or active infections requiring intravenous antimicrobials; symptomatic congestive heart failure defined as NYHA class III or IV; unstable angina pectoris within 6 months of study enrollment; history of myocardial infarction, stroke or intracranial hemorrhage within 6 months prior to enrollment; moderate to severe hepatic impairment (Child-Pugh class B or C); psychiatric illness or social situations that would limit compliance with study requirements
* Previous or current cancer, except curatively treated basal or squamous cell carcinoma of the skin, and curatively treated malignant melanoma stage 0-1A with a low risk of recurrence/metastasis as per assessment of the investigator, cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis and T1)
* Known HIV infection
* Infected with Hepatitis B or Hepatitis C viruses
* Participants with history of either untreated or inadequately treated latent or active TB infections/currently being treated for active TB
* Recent (within 21 days before visit 1) major surgery
* Participants who have history of a single episode of disseminated HZ or disseminated HS or recurrent (> 1 episode of) localized dermatomal HZ should be excluded
* Any gastrointestinal or metabolic condition that could interfere with the absorption of the oral medication
* History of thrombosis/thromboembolic event, known coagulopathy
* Have hearing loss with progression over the previous 5 years, sudden hearing loss, or middle or inner ear disease such as otitis media, cholesteatoma, Meniere's disease, labyrinthitis, or other auditory condition that is considered current, fluctuating, or progressive.
* Abnormality in hematology, chemistry profiles, or ECG during screening:

  * Platelet count: <100,000/ mm3
  * Lymphocytes: <600/ mm3
  * Absolute neutrophil count: <1200/ mm3
  * Hemoglobin: <9.0 g/dL
  * ALT or AST: >3.0xULN
  * eGFR: <30 mL/min
  * ECG that demonstrates clinically relevant abnormalities that may affect participant safety

Prior/Concomitant Therapy

* Less than 3 months have elapsed since last JAK inhibitors
* Glucocorticosteroids when used systematically within 1 month prior to visit 2
* Prior treatment with other concomitant investigational agents
* Hypersensitivity or allergic reaction to compounds related to JAK inhibitors
* Treatment with medication that might interfere with blood levels or have a major impact on the clinical readout of the study drug, as per discretion of the study investigator
* Participants who have received prohibited drugs that are CYP3A inducers within a 28 day or 5 half-lives (whichever is longer) period prior to the first dose of study intervention
* Participants who have received prohibited drugs that are CYP3A4 or CYP1A2 substrates with narrow therapeutic index where small concentration changes may lead to serious adverse reactions within 1 week or 5 half-lives (whichever is longer) period prior to the first dose of study intervention
* Participant has received a live attenuated vaccine ≤ 30 days prior to study screening
* Treatment with any anti-IgE therapies (eg, omalizumab, ligelizumab) within 1 months prior to screening visit

Other Exclusions

* Pregnant or breast-feeding women
* Unwillingness or inability to use a contraception method during the time of participation in the trial
* Active alcohol and/or drug abuse
* Participant is unable to complete a participant diary or complete questionnaires, or does not meet the required level of compliance (≥ 80%) with the diary

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Urticaria Activity Score (UAS7) | Baseline to Week 12
  The UAS7 is calculated by adding up the daily UAS scores over a 7-day period. The score ranges from 0 to 42, with higher scores indicating more active disease.
  Score Ranges:
  0: Urticaria-free; 1-6: Well-controlled urticaria; 7-15: Mild urticaria; 16-27: Moderate urticaria; 28-42: Severe urticaria.

SECONDARY OUTCOMES:
Change in Urticaria Activity Score (UAS7) | Baseline to Week 2, 4, 8, and 16
  The UAS7 is calculated by adding up the daily UAS scores over a 7-day period. The score ranges from 0 to 42, with higher scores indicating more active disease.
  Score Ranges:
  0: Urticaria-free; 1-6: Well-controlled urticaria; 7-15: Mild urticaria; 16-27: Moderate urticaria; 28-42: Severe urticaria.
Change in Angioedema Activity Score (AAS7) | Baseline to Week 2, 4, 8, and 16
  Questionnaire used to measure the severity of angioedema symptoms over a 7-day period, where patients rate different aspects of their angioedema experience on a scale, with a higher score indicating greater disease activity; it is often used to assess the effectiveness of treatments for angioedema conditions like chronic spontaneous urticaria (CSU) or chronic histaminergic angioedema (CHA). Each day, patients rate different aspects of their angioedema (duration, severity, impact on daily activities) on a scale from 0 to 3, and the daily scores are summed over 7 days to get the AAS7 score. The score ranges from 0 to 105, with higher scores indicating more severe angioedema activity. Low Score (0-6): Indicates minimal angioedema activity Moderate Score (7-18): Represents moderate angioedema activity High Score (19-105): Shows severe angioedema activity
Percentage change of Health-Related Quality of Life (CU-Q2oL) | Baseline to Week 12
  Survey that measures a patient's health-related quality of life (HR-QOL) in relation to chronic urticaria (CU). The CU-Q2oL is a 23-question survey that measures a patient's HR-QOL in relation to CU. The survey asks about a patient's sleep, concentration, energy levels, and how CU symptoms impact their daily life. The survey scores range from 1 (no complaints) to 5 (many complaints). which gives a total raw score from 0-115 which is then converted to provide Total score range from 0-100, with higher score indicating poorer health outcome.
Change in Urticaria Control Test (UCT) | Baseline to Week 12
  A 4 question survey with a 4 week recall to describe a patient's current health situation in relation to UC. Total score ranges from 0 -16, with higher score indicating better health outcomes. A score of 16 indicates complete disease control. A score of <12 on the UCT identifies patients with poorly controlled chronic urticaria (CU), and a score of ≥12 identifies those with well-controlled symptoms. An improvement in 3 points is a minimal response, and an improvement of ≥6 points is a marked response.
Percentage change in Urticaria Activity Score (UAS7) | Baseline to Week 2, 4, 8, 12, and 16
  The UAS7 is calculated by adding up the daily UAS scores over a 7-day period. The score ranges from 0 to 42, with higher scores indicating more active disease.
  Score Ranges:
  0: Urticaria-free; 1-6: Well-controlled urticaria; 7-15: Mild urticaria; 16-27: Moderate urticaria; 28-42: Severe urticaria.
Percentage change in Angioedema Activity Score (AAS7) | Baseline to Week 2, 4, 8, 12, and 16
  Questionnaire used to measure the severity of angioedema symptoms over a 7-day period, where patients rate different aspects of their angioedema experience on a scale, with a higher score indicating greater disease activity; it is often used to assess the effectiveness of treatments for angioedema conditions like chronic spontaneous urticaria (CSU) or chronic histaminergic angioedema (CHA). Each day, patients rate different aspects of their angioedema (duration, severity, impact on daily activities) on a scale from 0 to 3, and the daily scores are summed over 7 days to get the AAS7 score. Low Score (0-6): Indicates minimal angioedema activity Moderate Score (7-18): Represents moderate angioedema activity High Score (19-105): Shows severe angioedema activity
Percentage of participants achieving 80% or greater improvement in Urticaria Activity Score (UAS7) | Baseline to Week 12
  Percentage of participants achieving 80% or greater improvement in their weekly UAS7 score compare to baseline at week 12 and throughout the study. The UAS7 is calculated by adding up the daily UAS scores over a 7-day period. The score ranges from 0 to 42, with higher scores indicating more active disease.
  Score Ranges:
  0: Urticaria-free; 1-6: Well-controlled urticaria; 7-15: Mild urticaria; 16-27: Moderate urticaria; 28-42: Severe urticaria.
Percentage of participants with Response of Urticaria Activity | Baseline to Week 12
  Percentage of participants achieving complete response (CR: 100% improvement), partial response (PR: 50% to 99% reduction from the baseline UAS7 score), stable disease (SD: <25% increase to <50% clearance from baseline), and progressive disease (>25% worsening above the baseline score) in skin at week 12 and throughout the study.
Percentage Change in Cohort Response Rate of Urticaria Activity Score (UAS7) | Baseline to Week 12
  The UAS7 is calculated by adding up the daily UAS scores over a 7-day period. The score ranges from 0 to 42, with higher scores indicating more active disease.
  Score Ranges:
  0: Urticaria-free; 1-6: Well-controlled urticaria; 7-15: Mild urticaria; 16-27: Moderate urticaria; 28-42: Severe urticaria.

CONTACTS AND LOCATIONS:
Overall Officials: Ahuva Cices, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.